CLINICAL TRIAL: NCT04688788
Title: Danish Non-inferiority Study of Ocrelizumab and Rituximab in MS (DanNORMS): A Randomized Study Comparing the Efficacy of Ocrelizumab and Rituximab in Active Multiple Sclerosis
Brief Title: Non-inferiority Study of Ocrelizumab and Rituximab in Active Multiple Sclerosis
Acronym: DanNORMS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Odense University Hospital (Other); Aarhus University Hospital (Other); Aalborg University Hospital (Other); Herlev Hospital (Other); Hillerod Hospital, Denmark (Other); Kolding Sygehus (Other); Gødstrup Hospital (Other); Hvidovre University Hospital (Other); Hospital of South West Jutland, Esbjerg, Denmark (Unknown); GCP unit, Copenhagen University Hospital (Unknown); GCP-unit at Aarhus University Hospital, Aarhus, Denmark (Other); Hospital of Southern Jutland, Sønderborg, Denmark (Unknown); Hospital of Central Denmark Region, Viborg, Denmark (Unknown); Danske Regioner (Other); Hospital of Southern Jutland, Aabenraa, Denmark (Unknown); Sanquin Research & Blood Bank Divisions (Other)
Responsible Party: Principal Investigator, Jeppe Romme Christensen, National coordinating principal investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DanNORMS_version 3.2
Record Dates: First submitted 2020-12-22; First posted 2020-12-30 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Relapsing Remitting Multiple Sclerosis; Secondary Progressive Multiple Sclerosis; Primary Progressive Multiple Sclerosis
Keywords: Magnetic resonance imaging; Rituximab; Ocrelizumab
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive | interventions — Rituximab; ocrelizumab; fexofenadine; Acetaminophen; Methylprednisolone

STUDY DESIGN:
Intervention Model Description: A prospective, 2:1 randomized, open-label, multi-centre, phase 3 non-inferiority clinical trial with blinded primary endpoint.
Who Masked: Outcomes Assessor
Masking Description: MRI scan data will be transfered to the MRI Reader Centre with pseudonymized identity and without any information regarding the treatment allocation of the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rituximab (Experimental): Intravenous biosimilar rituximab (Ruxience®, Rixathon® or other biosimilar rituximab) 1000 mg given every 6th month (first 2 infusions 1000mg/1000 mg given 2 weeks apart).
  Interventions: Drug: Rituximab; Drug: Fexofenadine; Drug: Paracetamol; Drug: Methylprednisolone
- Ocrelizumab (Active Comparator): Intravenous ocrelizumab (Ocrevus®) 600 mg every 6th month (first 2 infusions 300 mg/300 mg given 2 weeks apart).
  Interventions: Drug: Ocrelizumab; Drug: Fexofenadine; Drug: Paracetamol; Drug: Methylprednisolone

INTERVENTIONS:
Drug: Rituximab — Rituximab is a chimeric mouse/human monoclonal immunoglobulin gamma-1 (IgG1) antibody which depletes cluster of differentiation antigen 20 (CD20)-positive cells. Rituximab is approved for non-hodgkin lymphoma, chronic lymphocytic leukemia, rheumatoid arthritis, granulomatosis with polyangitis and microscopic polyangitis, and pemphigus vulgaris.
  Other Names: Ruxience, Rixathon® or other biosimilar rituximab
  Arms: Rituximab
Drug: Ocrelizumab — Ocrelizumab is a recombinant humanised monoclonal IgG1 antibody which depletes CD20-positive cells. Ocrelizumab is approved for multiple sclerosis.
  Other Names: Ocrevus
  Arms: Ocrelizumab
Drug: Fexofenadine — Premedication with oral fexofenadine 360 mg is given before every infusion to reduce frequency and intensity of infusion related reactions.
Drug: Paracetamol — Premedication with oral. paracetamol 1000 mg is given before every infusion to reduce frequency and intensity of infusion related reactions.
Drug: Methylprednisolone — Premedication with oral methylprednisolone 100 mg is given before every infusion to reduce frequency and intensity of infusion related reactions.

SUMMARY:
The DanNORMS study is a phase 3, non-inferiority clinical trial examining whether treatment of active multiple sclerosis with rituximab is non-inferior to ocrelizumab regarding efficacy and safety.

DETAILED DESCRIPTION:
The DanNORMS study will include patients with active multiple sclerosis aged 18-65 years. Patients will be randomized in a 2:1 ratio to either rituximab or ocrelizumab. The study duration is 24 months for the core-phase, and patients can continue in a long-term follow-up phase for additional 36 months with possibility for extended interval dosing guided by CD19+ B cell count.

The primary endpoint is the percentage of patients without new or enlarging T2 white matter lesions on brain MRI scans from month 6 to month 24, which will be assessed by radiologists blinded to the treatments status. The study will evaluate a number of efficacy and safety endpoints using clinical, MRI, routine blood samples and research biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* MS diagnosis and definition of disease course according to the 2017 McDonald criteria
* Expanded disability status scale (EDSS) ≤6.5
* Fulfilling criteria for active MS:

  * Treatment naïve relapsing remitting multiple sclerosis (RRMS) patients (never treated, or no DMT the previous 2 years):

    1. ▪≥2 relapse previous 12 months OR
    2. 1 relapse previous 12 months with severe residual symptoms and EDSS ≥ 3.0 OR
    3. 1 relapse previous 12 months AND ≥9 T2 lesions on brain and/or spinal cord MRI AND

       * 1 contrast-enhancing lesion or ≥1 new or enlarging T2 lesion on brain and/or spinal cord MRI previous 12 month
  * Previously treated RRMS patients:

    1. ≥1 relapse previous 12 months OR
    2. ≥1 contrast-enhancing lesion or ≥2 new/enlarging T2 lesions on brain and/or spinal cord MRI previous 12 months
  * Progressive MS patients:

    1. ≥1 relapse previous 12 months OR
    2. ≥1 contrast-enhancing lesion previous 12 months or ≥1 new/enlarging T2 lesions on brain and/or spinal cord MRI previous 12 months or ≥2 new or enlarging T2 lesion on brain and/or spinal cord MRI previous 24 months OR
    3. Increased levels of neurofilament light chain (NFL) in serum or cerebrospinal fluid (CSF) in sample collected previous 12 months. Progressive MS patients not fulfilling the clinical/MRI criteria for active disease, may qualify for inclusion in the study if:

       (A) CSF NFL level (measured with NF-Light® ELISA assay from Uman Diagnostics or Simoa):
       * 18 to 40 years >560 ng/l
       * 41 to 60 years >890 ng/l
       * 61 to 65 years >1850 ng/l

       or

       (B) Serum NFL level (measured with Simoa™ NF-light® Advantage Kit)

       o Increased sNFL based on individual age-determined cut-off: >4.19 × 1.029^age ng/L

       OR

       o Increased sNFL based age-partitioned cut-offs:
       * 18 to 20 years >7.4 ng/L
       * 21 to 30 years >9.9 ng/L
       * 31 to 40 years >13.1 ng/L
       * 41 to 50 years >17.5 ng/L
       * 51 to 60 years >23.3 ng/L
       * 61 to 65 years >30.9 ng/L
* Signed written informed consent

Exclusion Criteria:

* Pregnancy or breast feeding
* Lack of effective contraception for women of child-bearing potential (effective contraception include oral contraception, intrauterine devices and other forms of contraception with failure rate <1%)
* Receipt of a live or live-attenuated vaccine within 6 weeks prior to randomization
* Known active malignant disease
* Severe heart failure (New York Heart Association Class IV) or severe, uncontrolled cardiac disease
* Positive test for HIV, hepatitis B or C, or symptoms or signs of active tuberculosis in a patient with a positive Quantiferon test.
* Negative test for varicella zoster
* Lymphopenia grade 2 (0.5 to 0.8 × 10^9/L) or higher grades of lymphopenia. In case of switching from fingolimod, siponimod or ozanimod lymphopenia is accepted at screening visit. Patients switching from dimethylfumarate who have persistent lymphopenia 5 to 6 weeks after stopping dimethylfumarate can be included if lymphopenia is grade 2 or lower, and treating phycisian judge CD20-depleting therapy safe.
* Neutropenia grade 2 (1.0 to 1.5 × 10^9/L) or higher grades
* Thrombocytopenia grade 2 (50 to 75 × 10^9/L) or higher grades
* Previous treatment with alemtuzumab or hematopoietic stem-cell transplantation
* Previous treatment with cladribine, CD20-depleting antibodies, daclizumab or other immune suppressive treatment which is judged to still exert immune suppressive effect by treating physician
* Methylprednisolone treatment within 1 month of baseline visit
* Findings on the screening MRI judged to preclude participation by the treating physician
* Other diseases judged to be relevant by the treating physician
* Contraindication to MRI
* Known allergy or hypersensitivity to rituximab or ocrelizumab

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2026-05-05 (Estimated); Study Completion 2029-05-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients without new or enlarging T2 white matter lesions on brain MRI scans | Month 6 to month 24
  MRI outcome

SECONDARY OUTCOMES:
Percentage of patients with 6-month confirmed disability progression (CDP) in Expanded Disability Status Scale (EDSS) | Baseline to month 24
  Clinical outcome
Annualised relapse rate based on cumulative number of confirmed relapses from baseline to months 24 | Baseline to month 24
  Clinical outcome
Percentage of patients with 6-months CDP in Timed 25 Foot Walk (T25FW) | Baseline to month 24
  Clinical outcome
Percentage of patients with 6-months CDP in 9-Hole-Peg Test (9HPT) | Baseline to month 24
  Clinical outcome
Percentage of patients with 6-months CDP in Symbol Digit Modalities Test (SDMT) | Baseline to month 24
  Clinical outcome
Change in Multiple Sclerosis Impact Scale (MSIS-29) | Baseline to month 24
  Patient related outcome measure (PROM). A 29 item questionnaire with values ranging from 29 (good) to 145 (worse).
Change in Fatigue Scale for Motor and Cognitive Functions (FSMC) | Baseline to month 24
  PROM. A 20 item questionnaire with values ranging from 20 (no fatigue at all) and 100 (severest grade of fatigue.
EuroQol- 5 Dimension (EQ-5D) | Baseline to month 24
  PROM. A 5 item questionnaire with values ranging from 5 (good) to 15 (worse).
Percentage of patients without gadolinium-enhancing lesions (GdEL) | Month 6 and month 24 MRI scans
  MRI outcome
Change in T2 white matter lesion volume | From month 6 to month 24
  MRI outcome
Change in T1 white matter lesion volume | From month 6 to month 24
  MRI outcome
Percentage brain volume change (PBVC) from month 6 to month 24 | From month 6 to month 24
  MRI outcome
Change in serum neurofilament light chain level | From baseline to month 24
  Blood biomarker
Blood levels of cluster of differentiation antigen 19 (CD19)+ B cells | At month 6 and month 24
  Blood biomarker

OTHER OUTCOMES:
Antidrug antibody frequency | Baseline, month 6 and month 24
  Anti drug antibodies against rituximab or ocrelizumab
Drug concentration | Month 6 and month 24
  Rituximab or ocrelizumab drug concentration
Genotyping of Fc gamma receptor type IIA and IIIA (FCRGIIA and FCGRIIIA), Complement C1q A Chain (C1QA) and low-density lipoprotein receptor-related protein 2 (LRP2) | Baseline
  Genotypes associated with rituximab efficacy and safety (FCRGIIA 131, FCGRIIIA 158, C1QA 276) and relapse frequency (LRP2)

CONTACTS AND LOCATIONS:
Overall Officials: Jeppe Romme Christensen, MD, PhD, Principal Investigator — Danish Multiple Sclerosis Center Rigshospitalet
Locations (11):
- Denmark (11):
  - Danish Multiple Sclerosis Center, Rigshospitalet, Glostrup Municipality, Copenhagen
  - Department of Neurology, Aalborg University Hospital, Aalborg
  - Department of Neurology, Aarhus University Hospital, Aarhus
  - Department of Neurology, Hospital of South West Jutland, Esbjerg, Esbjerg
  - Department of Neurology, Herlev Hospital, Herlev
  - Department of Neurology, Nordsjællands Hospital i Hillerød, Hillerød
  - Department of Neurology, Regionshospitalet Holstebro, Holstebro
  - Department of Neurology, Kolding Hospital, Kolding
  - Department of Neurology, Odense University Hospital, Odense
  - Department of Neurology, Hospital of Southern Jutland, Sønderborg, Sønderborg
  - Department of neurology, Regionshospitalet Viborg, Viborg

IPD SHARING:
Plan to Share IPD: No